CLINICAL TRIAL: NCT03181633
Title: An Open-Label Study to Evaluate Efficacy and Safety of Long-Term Treatment With ACH-0144471 in Participants Who Completed Clinical Study ACH471-100
Brief Title: A Long-Term Treatment Study of ACH-0144471 in Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH471-103; 2017-000665-79 (EudraCT Number); U1111-1196-0653 (Other: UTN)
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH; Paroxysmal; Hemoglobinuria; ACH-0144471; ALXN2040; Danicopan
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemoglobinuria | interventions — danicopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ACH-0144471 (Experimental): All participants will receive ACH-0144471 during the treatment period.
  Interventions: Drug: ACH-0144471

INTERVENTIONS:
Drug: ACH-0144471 — ACH-0144471 will be administered to all participants enrolled in the study.

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of ACH-0144471 in participants with paroxysmal nocturnal hemoglobinuria (PNH) who have demonstrated clinical benefit from ACH-0144471 in Study ACH471-100. This study is designed to include up to 12 participants.

ELIGIBILITY:
Inclusion Criteria:

* Study designed to include up to 12 participants who completed treatment in Study ACH471-100 and demonstrated clinical benefit from ACH-0144471 with no significant safety or tolerability concerns.
* Negative pregnancy test for females prior to dosing and throughout the study.

Exclusion Criteria:

* Have developed any clinically relevant co-morbidities while participating in Study ACH471-100 that would make the participant inappropriate for the continuation of treatment with ACH-0144471, in the opinion of the Investigator.
* Have developed any clinically significant laboratory abnormalities while participating in Study ACH471-100 that, in the opinion of the Investigator, would make the participant inappropriate for the study or put the participant at undue risk.
* Females who are pregnant, nursing, or planning to become pregnant during the study or within 90 days of study drug administration or participants with a female partner who is pregnant, nursing, or planning to become pregnant during the study or within 90 days of study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (2):
  - Clinical Trial Site, Avellino
  - Clinical Trial Site, Naples
- Clinical Trial Site, Auckland, New Zealand
- Clinical Trial Site, Seoul, South Korea

REFERENCES:
- [Derived] Kulasekararaj AG, Browett PJ, Risitano AM, Patriquin CJ, Yenerel MN, Marceau D, Sahin F, Algarra L, Ogawa M, Yu J, Cross N, Notaro R, Lee JW, Brodsky RA. Efficacy and Safety of Vemircopan as Monotherapy in Patients With Paroxysmal Nocturnal Hemoglobinuria. Blood Adv. 2025 Oct 22:bloodadvances.2025017731. doi: 10.1182/bloodadvances.2025017731. Online ahead of print. PMID 41124654

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who demonstrated a clinical benefit from danicopan in the primary Study ACH471-100 (NCT03053102), were eligible for long-term treatment with danicopan in this extension study ACH471-103.
Groups:
- Danicopan: Participants in this study continued to receive danicopan tablets orally at the same dose (150, 175, or 200 milligrams [mg] 3 times daily [TID]) that they were receiving upon completion of the primary Study ACH471-100. Dose escalation was done in increments of 25 mg to a maximum of 250 mg TID, in case additional clinical benefit was expected as per Investigator and Sponsor decision.
Period: Overall Study
Arm/Group | Danicopan
Started | 8
Received at Least 1 Dose of Study Drug | 8
Completed | 6
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Missing follow-up visit | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all enrolled and treated participants.
Arm/Group | Danicopan
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.51 (14.752)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 6
  Race: Asian | 1
  Race: Other | 1
Lactate Dehydrogenase (LDH) Level [Mean (Standard Deviation); unit: units (U)/liter (L)] | 1403.13 (602.824)
Hemoglobin (Hgb) Level in the Absence of Red Blood Cell (RBC) Transfusion [Mean (Standard Deviation); unit: grams (g)/liter (L)] | 96.50 (18.055)
Reticulocyte Counts [Mean (Standard Deviation); unit: 10^12 cells/L] | 0.15 (0.078)
Paroxysmal Nocturnal Hemoglobinuria (PNH) Clone Size [Mean (Standard Deviation); unit: percentage of the total cell population] — Population: Here, 'number analyzed' signifies participants evaluable for this baseline measure.
  percentage of the total cell population
    number analyzed (Participants) | 6
    (all) | 39.67 (29.696)
Free Hgb [Mean (Standard Deviation); unit: mg/deciliter (dL)] | 36.08 (42.417)
Alternative Pathway (AP) Complement Functional Activity [Mean (Standard Deviation); unit: percentage of activity] — Serum AP functional activity was measured by the Wieslab functional immunoassay method.
  percentage of activity | 66.70 (12.732)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in LDH Level at Week 25
Description: Change from Baseline = Serum LDH levels at Week 25 - Baseline Serum LDH levels. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Week 25
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the post baseline assessments for LDH level.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Danicopan
Number analyzed (Participants) | 7
U/L | -683.29 (845.175)

2. Primary Outcome: Change From Baseline in Hgb Level in the Absence of RBC Transfusion at Week 25
Description: Change from Baseline = Hgb levels at Week 25 - Baseline Hgb levels. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Week 25
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for Hgb level.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Danicopan
Number analyzed (Participants) | 6
g/L | 24.67 (18.052)

3. Primary Outcome: Change From Baseline in Reticulocyte Counts at Week 25
Description: Change from Baseline = reticulocyte count at Week 25 - Baseline reticulocyte count. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Week 25
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for reticulocyte count.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Danicopan
Number analyzed (Participants) | 7
10^12 cells/L | -0.07 (0.063)

4. Primary Outcome: Number of RBC Units Transfused
Time Frame: Baseline up to Week 169
Population: Full analysis set included all enrolled and treated participants.
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Danicopan
Number analyzed (Participants) | 8
RBC units | 6.5 (16.83)

5. Primary Outcome: Number of RBC Transfusion Instances
Time Frame: Baseline up to Week 169
Population: Full analysis set included all enrolled and treated participants.
Measure: Mean (Standard Deviation); unit: RBC transfusion instances
Arm/Group | Danicopan
Number analyzed (Participants) | 8
RBC transfusion instances | 3.4 (8.00)

6. Primary Outcome: Change From Baseline in PNH Clone Size at Week 25
Description: The PNH clone size refers to the percentage of PNH-affected cells versus normal cells within the total cell population. Change from Baseline = PNH clone size at Week 25 - Baseline PNH clone size. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Week 25
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for PNH clone size.
Measure: Mean (Standard Deviation); unit: percentage of the total cell population
Arm/Group | Danicopan
Number analyzed (Participants) | 5
percentage of the total cell population | 22.00 (5.831)

7. Primary Outcome: Change From Baseline in AP Complement Functional Activity at Week 25
Description: Serum AP functional activity was measured by the Wieslab functional immunoassay method. Change from Baseline = Serum AP functional activity at Week 25 - Baseline Serum AP functional activity. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Week 25
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for Serum AP functional activity.
Measure: Mean (Standard Deviation); unit: percentage of activity
Arm/Group | Danicopan
Number analyzed (Participants) | 7
percentage of activity | -46.36 (25.316)

8. Primary Outcome: Change From Baseline in Free Hgb at Week 25
Description: Change from Baseline = free Hgb at Week 25 - Baseline free Hgb. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Week 25
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for free Hgb.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Danicopan
Number analyzed (Participants) | 6
mg/dL | 59.83 (66.414)

9. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Grade 3 and Grade 4 Adverse Events (AEs), And AEs Leading To Discontinuation
Description: An AE was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. The intensity of an AE was graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Adverse Event Severity Grading Table. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to 4.5 years
Population: Safety analysis set included all enrolled participants who received at least 1 dose of danicopan.
Measure: Number; unit: participants
Arm/Group | Danicopan
Number analyzed (Participants) | 8
participants
  Any TEAEs | 8
  SAEs | 3
  TEAE Grade 3 | 2
  TEAE Grade 4 | 0
  AE leading to discontinuation | 0

10. Secondary Outcome: Change From Baseline in LDH Level at Weeks 49 and 169
Description: Change from Baseline = Serum LDH levels at specified postbaseline visit - Baseline Serum LDH levels. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Weeks 49 and 169
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for LDH level. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Danicopan
Number analyzed (Participants) | 6
U/L
  Change at Week 49 | -862.50 (568.302)
  Change at Week 169: number analyzed (Participants) | 2
  Change at Week 169 | -1388.00 (562.857)

11. Secondary Outcome: Change From Baseline in Hgb Level in the Absence of RBC Transfusion at Weeks 49 and 169
Description: Change from Baseline = Hgb levels at specified postbaseline visit - Baseline Hgb levels. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Weeks 49 and 169
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for Hgb level. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Danicopan
Number analyzed (Participants) | 5
g/L
  Change at Week 49 | 21.40 (18.995)
  Change at Week 169: number analyzed (Participants) | 2
  Change at Week 169 | 54.50 (14.849)

12. Secondary Outcome: Change From Baseline in Reticulocyte Counts at Weeks 49 and 169
Description: Change from Baseline = reticulocyte count at specified postbaseline visit - Baseline reticulocyte count. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Weeks 49 and 169
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for reticulocyte count. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Danicopan
Number analyzed (Participants) | 6
10^12 cells/L
  Change at Week 49 | -0.05 (0.065)
  Change at Week 169: number analyzed (Participants) | 2
  Change at Week 169 | -0.12 (0.049)

13. Secondary Outcome: Change From Baseline in PNH Clone Size at Weeks 49 and 73
Description: The PNH clone size refers to the percentage of PNH-affected cells versus normal cells within the total cell population. Change from Baseline = PNH clone size at specified postbaseline visit - Baseline PNH clone size. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Weeks 49 and 73
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for PNH clone size. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of the total cell population
Arm/Group | Danicopan
Number analyzed (Participants) | 6
percentage of the total cell population
  Change at Week 49 | 30.83 (11.531)
  Change at Week 73: number analyzed (Participants) | 5
  Change at Week 73 | 32.00 (19.170)

14. Secondary Outcome: Change From Baseline in AP Complement Functional Activity at Weeks 49 and 145
Description: Serum AP functional activity was measured by the Wieslab functional immunoassay method. Change from Baseline = Serum AP functional activity at specified postbaseline visit - Baseline Serum AP functional activity. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Weeks 49 and 145
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for Serum AP functional activity. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of activity
Arm/Group | Danicopan
Number analyzed (Participants) | 6
percentage of activity
  Change at Week 49 | -59.80 (14.217)
  Change at Week 145: number analyzed (Participants) | 2
  Change at Week 145 | -52.43 (2.779)

15. Secondary Outcome: Change From Baseline in Free Hgb at Weeks 49 and 169
Description: Change from Baseline = free Hgb at specified postbaseline visit - Baseline free Hgb. Baseline was the baseline value from the primary Study ACH471-100.
Time Frame: Baseline, Weeks 49 and 169
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for free Hgb. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Danicopan
Number analyzed (Participants) | 6
mg/dL
  Change at Week 49 | 105.92 (92.308)
  Change at Week 169: number analyzed (Participants) | 2
  Change at Week 169 | -30.75 (54.942)

16. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Score at Weeks 21, 41, and 153
Description: The FACIT-Fatigue scale is a collection of quality of life questionnaires pertaining to the management of fatigue symptoms due to a chronic illness. The FACIT-Fatigue is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the preceding 7 days. Participants score each item on a 5-point scale: 0 (Not at all) to 4 (Very much). Total scores range from 0 to 52, with higher score indicating better quality of life.
Time Frame: Baseline, Weeks 21, 41, and 153
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for FACIT-Fatigue scale score. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Danicopan
Number analyzed (Participants) | 8
units on a scale
  Change at Week 21 | 8.4 (11.75)
  Change at Week 41: number analyzed (Participants) | 7
  Change at Week 41 | 9.1 (13.37)
  Change at Week 153: number analyzed (Participants) | 2
  Change at Week 153 | 3.0 (0.00)

17. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire-Core 30 Scale (EORTC-QLQ-C30): Global Health Status/Qol Score at Weeks 21, 41, and 153
Description: EORTC-QLQ-C30 is comprised of 30 questions. First 28 questions used 4-point scale (1=not at all,2=a little,3=quite a bit,4=very much) for evaluating 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (fatigue, nausea/vomiting, pain) & other single items. For each item, high score = high level of symptomatology/problem. Last 2 questions represented participant's assessment of overall health (global health status) and quality of life, coded on 7-point scale (1=very poor to 7=excellent). Answers were converted into grading scale, with total score between 0 and 100. A high score represented a favourable outcome with a best quality of life for participant.
Time Frame: Baseline, Weeks 21, 41, and 153
Population: Full analysis set included all enrolled and treated participants. Here, 'Overall number of participants analyzed' = participants with both baseline and the postbaseline assessments for EORTC-QLQ-C30 (Global Health Status/Qol) score. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Danicopan
Number analyzed (Participants) | 8
units on a scale
  Change at Week 21 | 16.67 (25.973)
  Change at Week 41: number analyzed (Participants) | 7
  Change at Week 41 | 11.90 (29.603)
  Change at Week 153: number analyzed (Participants) | 2
  Change at Week 153 | 4.17 (17.678)

ADVERSE EVENTS:
Time Frame: Baseline up to 4.5 years
Description: Safety analysis set included all enrolled participants who received at least 1 dose of danicopan.
Arm/Group | Danicopan
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Danicopan (N=8)
Cystitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Haemolysis (Blood and lymphatic system disorders) | 1
Pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Danicopan (N=8)
Dysphagia (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 3
Pyrexia (General disorders) | 3
Fatigue (General disorders) | 1
Chest discomfort (General disorders) | 1
Influenza like illness (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Headache (Nervous system disorders) | 3
Lethargy (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Haemoglobinuria (Renal and urinary disorders) | 2
Chromaturia (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Haemolysis (Blood and lymphatic system disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT03181633/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT03181633/SAP_001.pdf